CLINICAL TRIAL: NCT01450436
Title: Impact of Preterm Body Composition at Discharge on 2 Years Neurological Development (ASQ Evaluation)
Acronym: EPIPOD
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROG/11/80
Record Dates: First submitted 2011-09-28; First posted 2011-10-12 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Other Preterm Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- preterm infants (<35 weeks gestation)
  Interventions: Other: Peapod assessment

INTERVENTIONS:
Other: Peapod assessment — EPIPOD consists in a Non-Interventional Research according to French regulations. Actually, Peapod examination at discharge takes part of current clinical practice and patient management in Nantes Neonatal Intensive Care Unit since 2008.
  After checking inclusion and non-inclusion criteria and obtaining oral informed consent from newborn legal authority or parents, PEAPOD assessment was leaded in the last week of hospitalization. Consisting in 2 repeated measurement, body composition estimation was completed by clinical and demographic data as neonatal nutrition (Parenteral nutrition pattern at Day 5, 10 and 21, and ASQ/BLR Neurodevelopmental assessment at 2 years old).

SUMMARY:
Neonatal nutritional management consists in reproducing miming uteri growth kinetic. Since the seventies, NICU (Neonatal Intensive Care Unit) strategy consists in a high proteidic input (apport) supposed to allow optimal neurodevelopment. However, nutritional practices and strategies have significantly evolved during these last years, influenced by Baker nutritional imprinting concept (2002). Actually, neonatal high proteidic exposition could perturb metabolism and hormonal systems of newborns conducting to a reinforcement of obesity and cardio-vascular pathology prevalence in this target population at adulthood. In this context many studies emerged since 2000 and try to assess the trade-off between neurodevelopment and growth under nutrition conditions. EPIPOD try to focus the link between heterogenous proteic input dispensed in our NICU (described by tercil methods on population) and fat mass phenotype variations at discharge (described by tercil methods); and its consequences on neurodevelopmental growth. Understanding how particular nutritional exposition could determine "fatty" phenotype and impact neurodevelopment is clearly our main goal.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns (< 35 weeks gestation).
* Final clinical discharge (No transfer)
* Oral Parental consent.
* Nantes NICU Neonatal management in the first 5 days of life

Exclusion Criteria:

* Congenital pathology inconsistent with PEAPOD investigation (Beckwith-Wiedemann syndrome, lipodystrophia with abnormal constitutional fat mass level).
* Pathology inducing neurodevelopment troubles.
* Transfer in an other hospital before discharge
* Hemodynamic or cardiovascular instability requiring continuous monitoring or perfusion, incompatible with PEAPOD measurement

Ages: 25 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants (< 35 weeks gestation)
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Fatty mass percentage at discharge by PEAPOD measurement | PEAPOD measurement will be done at newborns discharge, at an expected average of 6.4 weeks hospitalization
  After checking inclusion and non-inclusion criteria and obtaining oral informed consent from newborn legal authority or parents, PEAPOD assessment was leaded in the last week of hospitalization. Consisting in 2 repeated measurement, body composition estimation was completed by clinical and demographic data as neonatal nutrition (Parenteral nutrition pattern at Day 5, 10 and 21, and ASQ/BLR Neurodevelopmental assesmment at 2 years old).
Children neurological development at 2 years old evaluated by Ages and stages questionnaires (ASQ) | ASQ/BLR Neurodevelopmental assesmment at 2 years old.

SECONDARY OUTCOMES:
body composition of preterm infants at discharge and full term newborns at 3 days of life | PEAPOD measurement will be done at newborns discharge, at an expected average of 6.4 weeks hospitalization
Relationship between body composition at discharge and that at 2 years | PEAPOD measurement will be done at newborns discharge, at an expected average of 6.4 weeks hospitalization
Impact of fatty mass percentage at preterm newborns discharge on neurologic outcome assessed by a revised Brunet-Lezine test at 2 years. | PEAPOD measurement will be done at newborns discharge, at an expected average of 6.4 weeks hospitalization
Preterm infants feeding behavior at 2 years | At 2 years old
Factors (both intrinsic and nutritional) influencing body composition of preterm infants (<35 weeks gestation), at discharge | factors influencing body composition report will be done at newborns discharge, at an expected average of 6.4 weeks hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: FRONDAS-CHAUTY Anne, MD, Study Director — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Simon L, Frondas-Chauty A, Senterre T, Flamant C, Darmaun D, Roze JC. Determinants of body composition in preterm infants at the time of hospital discharge. Am J Clin Nutr. 2014 Jul;100(1):98-104. doi: 10.3945/ajcn.113.080945. Epub 2014 May 7. PMID 24808483